CLINICAL TRIAL: NCT02559674
Title: Phase Ib/II Study of ALT-803 in Combination With Gemcitabine and Nab-paclitaxel in Patients With Advanced Pancreatic Cancer
Brief Title: QUILT-2.001: ALT-803 in Patients With Advanced Pancreatic Cancer in Conjunction With Gemcitabine and Nab-Paclitaxel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altor BioScience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-ALT-803-01-15
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Advanced Pancreatic Cancer
Keywords: Pancreas; Pancreatic; Cancer; Advanced Pancreatic Cancer; Immunotherapy; Immunotherapeutic; Interleukin-15; Gemcitabine; Nab-paclitaxel; Solid Tumor; Metastatic Disease; Combination Immunotherapy
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phase Ib/II ALT-803 w/ gemcitabine and nab-paclitaxel (Experimental)
  Interventions: Biological: Gemcitabine; Biological: Nab-paclitaxel; Biological: ALT-803

INTERVENTIONS:
Biological: Gemcitabine — Intravenous Infusion; Patients will receive two 4-week treatment cycles consisting of gemcitabine given on Day 1, 8, 15, 29, 36, and 43. Eligible patients may receive up to 10 additional treatment cycles.
  Other Names: Gemzar
Biological: Nab-paclitaxel — Intravenous Infusion; Patients will receive two 4-week treatment cycles consisting of nab-paclitaxel given on Day 1, 8, 15, 29, 36, and 43. Eligible patients may receive up to 10 additional treatment cycles.
  Other Names: Abraxane
Biological: ALT-803 — Subcutaneous Injection; Patients will receive two 4-week cycles consisting of ALT-803 given on Day 2, 9, 16, 30, 37, and 44. Eligible patients may receive up to 10 additional treatment cycles.

SUMMARY:
This is a Phase Ib/II, open-label, multi-center, competitive enrollment and dose escalation study of ALT-803 in combination with gemcitabine and nab-paclitaxel in patients with advanced pancreatic cancer in conjunction with gemcitabine and nab-paclitaxel.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability of escalating doses, to identify the Maximum Tolerated Dose (MTD) and designate a dose level for Phase II study (RP2D) of ALT-803 administered in combination with gemcitabine and nab-paclitaxel in patients with advanced pancreatic cancer.

To access the anti-tumor activity of ALT-803 administered in combination with gemcitabine and nab-paclitaxel as measured by objective response rate, overall survival, progression-free survival, time to progression, and duration of response in patients with advanced pancreatic cancer.

To Characterize the pharmacokinetic, immunogenicity, and serum cytokine profile of ALT-803 in combination with gemcitabine and nab-paclitaxel in treated patients. To correlate circulating cell free DNA and circulating tumor DNA with clinical outcomes of the study in treated patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of pancreatic cancer.

  * For dose escalation phase (Phase Ib) distant metastatic disease or unresectable disease and not a candidate for down staging to resection.
  * For expansion phase (Phase II) distant metastatic disease only.
* For dose escalation phase (Phase Ib) 0 or 1 prior lines of chemotherapy for advanced pancreatic cancer. Prior gemcitabine is allowed, however prior nab-paclitaxel is not allowed.
* For expansion phase (Phase II) no prior therapy for pancreatic cancer is allowed except for adjuvant therapy as long as it was completed ≥ 6 months prior to study treatment start
* Have at least one untreated and progressing tumor lesion that can be accurately measured according to Response Evaluation Criteria in Solid Tumor
* Prior radiation is allowed if the index lesion(s) remains outside of the treatment field or has progressed since prior treatment. Radiation therapy must have been completed at least 4 weeks prior to the baseline scan
* Resolved acute effects of any prior therapy to baseline or Grade ≤1
* The Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2
* Life expectancy ≥12 weeks
* Glomerular Filtration Rate (GFR) > 40mL (milliliter)/min; Creatinine ≤ 1.5 x ULN (Upper limit of Normal)
* Platelets ≥100,000/uL (microliter)
* Hemoglobin ≥ 9g/dL
* Absolute Lymphocytes ≥800/uL
* Absolute neutrophil count/absolute granulocyte count ≥1500/uL
* Total bilirubin ≤ 2.0 X ULN, or ≤ 3.0 X ULN (for patients with Gilbert's Syndrome)
* aspartate aminotransferase, alanine aminotransferase ≤ 2.5 X ULN, or ≤ 5.0 X ULN (if liver metastasis present)
* Normal clinical assessment of pulmonary function
* Negative serum pregnancy test if female and of childbearing potential
* Subjects, both females and males, with reproductive potential must agree to use effective contraceptive measures for the duration of the study
* Must provide informed consent and HIPPA authorization and agree to comply with all protocol-specified procedures and follow-up evaluations

Exclusion Criteria:

* No women who are pregnant or nursing
* No known hypersensitivity to gemcitabine or nab-paclitaxel
* No concurrent herbal or unconventional therapy
* No prior therapy with IL-15 or IL-15 analog
* No ongoing toxicity from prior anti-cancer treatment that may interfere with study treatment. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must resolve to grade 1 or baseline before administration of the study treatment.
* No positive Hep C serology or active Hep B infection
* No congestive heart failure < 6 months
* No unstable angina pectoris < 6 months
* No myocardial infarction < 6 months
* No history of ventricular arrhythmias or severe cardiac dysfunction
* No history of uncontrollable supraventricular arrhythmias
* No New York Heart Association Class > II congestive heart failure
* No marked baseline prolongation of QT/QTc interval
* No known autoimmune disease requiring active treatment. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment. Inhaled or topical steroids, and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* No known prior organ allograft or allogeneic transplantation
* No known HIV-positive or AIDS unless patient is on a stable highly active antiretroviral therapy (HAART) regimen, have CD4 (cluster of differentiation 4) counts >350, with no detectable viral load on quantitative polymerase chain reaction test
* No untreated central nervous system metastases, or if treated must be neurologically stable for at least 2 weeks prior to enrollment
* No corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent)
* No psychiatric illness/social situation that would limit compliance
* No other illness that in the opinion of the investigator would exclude the subject from participating in the study
* No active systemic infection requiring parenteral antibiotic therapy
* No anti-cancer treatment including surgery, radiotherapy, chemotherapy, other immunotherapy, or investigational therapy within 14 days before treatment start
* No disease requiring systemic immunosuppressive therapy
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 3 years after surgical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07; Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
Determination of MTD; Phase Ib | 9 Months
  Determine the maximum tolerated dose (MTD) level and designate the recommended dose level for phase II.
Safety Profile (Number and severity of treatment related AEs); Phase Ib and II | 48 Months
  Number and severity of treatment related adverse events (AEs) that occur or worsen after the first dose of study treatment
Overall Survival; Phase II | 8.5 Months
  Determine the 8.5 month overall survival of treated patients

SECONDARY OUTCOMES:
Objective response rate | 72 Months
  Evaluate objective response rate in treated patients.
Duration of response | 72 Months
  Evaluate duration of response in treated patients.
Time to progression | 72 Months
  Evaluate time to progression in treated patients.
Progression-free survival | 72 Months
  Evaluate progression-free survival in treated patients.
Biomarkers; Phase Ib | 36 Months
  Measure the serum levels of the following including but not limited to Interleukin-2 (IL-2), Interleukin-4 (IL-4), Interleukin-6 (IL-6), Interleukin-10 (IL-10), Interferon-gamma (IFN-ɣ), Tumor necrosis factor-alpha (TNF-α) and Monocyte chemoattractant protein-1 (MCP-1)
Determine the level of anti-ALT-803 antibodies in patient serum | 36 Months
  Determine the level of anti-ALT-803 antibodies in patient serum
Area under the plasma concentration-time curve from time zero to infinity (AUC); Phase Ib | 36 Months
  Area under the plasma concentration-time curve from time zero to infinity (AUC)
Correlation between the level of circulating cell free DNA in patient plasma and response to study treatment | 36 Months
  Correlation between the level of circulating cell free DNA in patient plasma and response to study treatment
Correlation between the level of tumor DNA in patient plasma and response to study treatment | 36 Months
  Correlation between the level of tumor DNA in patient plasma and response to study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hing C. Wong, Ph.D., Study Chair — Altor BioScience
Locations (1):
- University of Hawaii Cancer Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No